CLINICAL TRIAL: NCT05029557
Title: The Effect of Education and Telephone Follow-up Based on the Chronic Care Model on Self-efficacy and Patient-reported Outcomes in COPD Patients
Brief Title: The Effect of Education Based on the Chronic Care Model in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Yasemin SAZAK, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HasanKU-SAZAK-001
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Self-Management; Nursing Care
Keywords: Chronic Care Model
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group patients (No Intervention): The patients in the Control Group will continue their routine procedures.
- Education and telephone follow ups based on the Chronic Care Model (Experimental): Intervention Group will be given training (0 months) with the training booklet, which is prepared by the researcher based on the Chronic Care Model, and which includes information and suggestions about self-management strategies. The training will be organized in one single session in a way not to exceed approximately 45-50 minutes. The patients, who will be included in the Intervention Group, will be followed up by phone every two weeks. Also, reminders and informative information based on the training booklet will be sent to patients every week in the form of a short message.
  Interventions: Behavioral: Education and telephone follow ups based on the Chronic Care Model

INTERVENTIONS:
Behavioral: Education and telephone follow ups based on the Chronic Care Model — The effects of Chronic Care Model-based education and telephone follow-up given to patients with COPD on self-efficacy and patient-reported outcomes.
  Arms: Education and telephone follow ups based on the Chronic Care Model

SUMMARY:
Individuals who have COPD need a nursing service, which provides qualified and effective professional care, self-care, and supportive care to perform their daily life activities, and improve their quality of life. It is predicted that the Chronic Care-Based Training Program to be implemented and the follow-ups can increase the level of self-efficacy and satisfaction, and raise awareness on the management of the disease in patients. The purpose of the study was to evaluate the effects of the Chronic Care Model based education and telephone follow-up given to patients with COPD on self-efficacy and patient-reported outcomes. Also, the Modified Patient-Reported Outcome Scale for Chronic Obstructive Pulmonary Disease-mCOPD-PRO scale, which will be used in the study, will be adapted into Turkish language and culture, and will be used in the study after its validity and reliability are examined.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease is a major global healthcare problem with its high prevalence, increasing incidence (partly due to population aging), and major serious personal, social, and economic costs. Individuals who have COPD require a nursing service that provides qualified and effective professional care, self-care, and supportive care to perform their daily life activities and improve their quality of life. Nurses have active roles in the management of COPD as professional members of the team, and perform the roles of caregiving, consultancy, researcher, manager, and trainer in COPD management. The skills needed for the management of COPD and the knowledge and interventions to develop these skills are conceptualized as self-management, which is a complex structure including drug compliance, smoking cessation, maintaining and increasing exercise capacity, healthy lifestyle changes that include nutrition regulation, vaccination, and symptom management. The purpose of "Self-management" in COPD is stated in the GOLD 2021 report as "to provide motivation, encouragement, and guidance for patients to acquire positive health behaviors and to gain the ability to cope with their disease". The Self-Management Training and Guidance provided by healthcare staff must be the basic element of the "Chronic Diseases Care Model" in the scope of the healthcare provided. Although various models were proposed for chronic disease management, the best known, most used, and most effective among these is the Chronic Care Model. The model has the quality of being a roadmap for high-quality and patient-centered service delivery in chronic diseases. Four components of the Chronic Care Model will be implemented in the present study, which are; Decision Making Support, Self-Management Support, Health Services Delivery Plan, and Clinical Information Systems. The study has a randomized controlled experimental study design. The sampling of the study will consist of the patients who were diagnosed with COPD, hospitalized in Elbistan State Hospital Chest Policlinic of Kahramanmaraş Provincial Health Directorate, met the inclusion criteria, and who volunteer to participate in the study. A total of 66 patients, 33 in the Control Group, and 33 in the Intervention Group will be randomized into groups in the computer medium.

According to the intervention protocol of the study,

1. A training booklet will be created for COPD patients in the scope of the Chronic Care Model self-management support component of the study. The quality of the booklet will be evaluated by submitting it to expert opinions.
2. Patients who meet the inclusion criteria will be included in the present study as the Intervention and Control Group according to the randomization list.
3. Patients in the Control and Intervention Group will be interviewed and their pre-test data will be collected after informed consent is obtained from them. For this purpose, Patient Information Form, COPD Self-Efficacy Scale, 6MWT, COPD Assessment Test (CAT),modified Medical Research Council (mMRC) Dyspnea Scale, Modified Patient-Reported Outcome Scale for Chronic Obstructive Pulmonary Disease (mCOPD-PRO) Scale will be used.
4. After the pre-tests are completed, the patients in the Intervention Group will be given training (0 months) with the training booklet, which is prepared by the researcher based on the Chronic Care Model, and which includes information and suggestions about self-management strategies. The training will be organized in one single session in a way not to exceed approximately 45-50 minutes.
5. The patients, who will be included in the Intervention Group, will be followed up by phone every two weeks. Also, reminders and informative information based on the training booklet will be sent to patients every week in the form of a short message.
6. The patients in the Control Group will continue their routine procedures.
7. Post-tests will be applied to the patients who will be included in the Control and Intervention Group at the 3rd-month polyclinic follow-up. The Patient Assessment of Chronic Illness Care (PACIC) will be used in this post-test in addition to the pre-tests. At the end of the study, Training will be given to the Control Group patients along with Training Booklet.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Confirmed COPD diagnosis
* Ability to communicate and literate
* Able to communicate by phone
* Volunteering to participate in the research.

Exclusion Criteria:

* Being closed to communication
* Unable to communicate by phone
* Not being a volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of self-efficacy status | 0 months
  The COPD Self-Efficacy Scale consists of 34 items and 5 subscales, and is used to determine the degree of confidence of COPD patients in managing or avoiding breathing difficulties in certain activities. The sub-factors of the scale consist of negative impact, emotional state, physical effort, weather/environment effect, and behavioral risk factors. On the scale, as the mean score increases, the degree of confidence also increases in managing or avoiding respiratory distress.
Evaluation of self-efficacy status | 3 months
  The COPD Self-Efficacy Scale consists of 34 items and 5 subscales, and is used to determine the degree of confidence of COPD patients in managing or avoiding breathing difficulties in certain activities. The sub-factors of the scale consist of negative impact, emotional state, physical effort, weather/environment effect, and behavioral risk factors. On the scale, as the mean score increases, the degree of confidence also increases in managing or avoiding respiratory distress.
Evaluation of patient-reported results | 0 months
  Modified Patient-Reported Outcome Scale for Chronic Obstructive Pulmonary Disease-mCOPD-PRO; The Turkish version of the scale will be used in the research after being adapted to the Turkish language and culture and examining its validity and reliability by the researcher. The scale consists of 27 items and physiological (17 items), psychological (7 items), and environmental (3 items) fields. The mCOPD-PRO is not a mere measurement of symptoms, it is a comprehensive measurement of disease-specific health status including physiological, psychological, and environmental domains. Each item consists of a 5-point Likert-type design, and the scores of the scale are graded between 0-4.
Evaluation of patient-reported results | 3 months
  Modified Patient-Reported Outcome Scale for Chronic Obstructive Pulmonary Disease-mCOPD-PRO; The Turkish version of the scale will be used in the research after being adapted to the Turkish language and culture and examining its validity and reliability by the researcher. The scale consists of 27 items and physiological (17 items), psychological (7 items), and environmental (3 items) fields. The mCOPD-PRO is not a mere measurement of symptoms, it is a comprehensive measurement of disease-specific health status including physiological, psychological, and environmental domains. Each item consists of a 5-point Likert-type design, and the scores of the scale are graded between 0-4.

SECONDARY OUTCOMES:
The Patient Assessment of Chronic Illness Care | 3 months
  The Patient Assessment of Chronic Illness Care (PACIC) is a relatively brief 20-item questionnaire designed to assess the extent to which care is aligned with the Chronic Care Model. It consists five factors and, 20-item. The increase in the scale scores shows that individuals with chronic disease are highly satisfied with the care they receive.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin OLGUN, Professor, Study Director — Hasan Kalyoncu University Faculty of Nursing
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sazak Y, Olgun N. The effect of Chronic Care Model-based follow-up on self-efficacy and patient-reported outcomes in COPD patients: a randomized controlled study. BMC Nurs. 2025 May 22;24(1):578. doi: 10.1186/s12912-025-03247-x. PMID 40405196